CLINICAL TRIAL: NCT06355479
Title: A Phase 3 Randomized, Double-blind, Active-controlled Multi-center Study to Evaluate the Efficacy, Safety of OsrHSA in Patients of Hepatic Cirrhosis With Hypoalbuminemia
Brief Title: A Study to Evaluate the Efficacy and Safety of OsrHSA in Patients of Hepatic Cirrhosis With Hypoalbuminemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Healthgen Biotechnology Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HY1001-2022-P3
Record Dates: First submitted 2024-03-21; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Hypoalbuminemia; Hepatic Cirrhosis
MeSH Terms: conditions — Hypoalbuminemia; Liver Cirrhosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- OsrHSA (Experimental): OsrHSA 20g, IV qd, Day1 up to Day 14
  Interventions: Drug: OsrHSA
- pHSA (Active Comparator): pHSA 20g, IV qd, Day1 up to Day 14
  Interventions: Drug: Plasbumin®-20

INTERVENTIONS:
Drug: OsrHSA — Recombinant Human Serum Albumin from Oryza Sativa
  Arms: OsrHSA
Drug: Plasbumin®-20 — Albumin (Human) 20%, USP
  Arms: pHSA

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of OsrHSA works to treat hypoalbuminemia in hepatic cirrhosis patients. It will also learn about the safety and immunogenicity of OsrHSA. The main question it aims to answer is whether OsrHSA is effective in elevating the serum albumin level of cirrhotic patients with hypoalbuminemia.

Researchers will compare OsrHSA to the positive comparator, plasma-derived HSA (pHSA) to see if OsrHSA presents as non-inferior to pHSA in the indication of hypoalbuminemia in hepatic cirrhosis patients.

Participants will be randomized in a 1:1 ratio to receive OsrHSA or HpHSA (20g IV qd) for up to 14 days, following an EOT visit. Follow-up visits will be taken on EOT+7d, EOT+14d, and EOT+30d, respectively.

ELIGIBILITY:
Main Inclusion Criteria:

1. Diagnosis of hepatic cirrhosis
2. Adult males or females, aged 18-75 years (both inclusive) at the time of consent
3. Serum albumin level ≤ 30 g/L
4. Capable of giving informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form and this protocol

Main Exclusion Criteria:

1. History of allergy to rice; a history of allergy to any component of the HpHSA product
2. Therapeutic/ Large-volume paracentesis (> 5L each time) during the treatment period
3. Ascites resulted from non-hepatic cirrhosis, Budd-Chiari syndrome
4. Participants with Grade III or Grade IV hepatic encephalopathy using West Heaven Criteria
5. A transjugular intrahepatic peritoneal shunt (TIPS) is performed within 1 month prior to the first dosing
6. Evidence of upper gastrointestinal hemorrhage 6 months prior to the first dosing
7. Participants with stage C and stage D hepatocellular carcinoma according to China Liver Cancer Staging (CNLC) Classification
8. Evidence of extrahepatic neoplastic disorders
9. Transplantation
10. HIV positive
11. Participants with pleural effusion and need therapeutic thoracentesis during the treatment period
12. Uncontrolled infection with body temperature ≥ 38.5 degrees Celsius (101.3 degrees Fahrenheit) or ≤ 35 degrees Celsius (95 degrees Fahrenheit) and white blood cells > 12.0×10^9/L. i.e. severe intraabdominal infections, sepsis, respiratory tract infections, urine tract infections.
13. Other serious underlying diseases, including but not limited to: hepatopulmonary syndrome, heart failure grade III-IV (NYHA scale of heart function), severe structural heart disease, symptomatic ischemic heart disease, severe chest and lung disease, hemodialysis, active biliary obstructive disease, etc.
14. With the following abnormal laboratory test values:

    Hematology: white blood cell count < 2.0×10^9/L, absolute neutrophil count < 1.0×10^9/L, platelets < 30×10^9/L, or hemoglobin < 75 g/L; Chemistry: ALT and/or AST > 5× upper limit of normal (ULN), total bilirubin > 3× ULN; Coagulation: INR>2.0; Renal function: Cr > 2×ULN, urine protein >2+; Echocardiography: LVEF < 50%
15. Pregnant or breastfeeding or plan to get pregnant in 6 months
16. Potentially fertile participants (other than women who have undergone hysterectomy, bilateral salpingectomy, bilateral tubal ligation, or postmenopause for more than 1 year, and men who have undergone bilateral vasectomy) who do not consent to or are unable to use effective contraception throughout the study and 120 days after the end of the study (or early discontinuation of the study);
17. Enrolled in any clinical trials within 3 months prior to the first dose of study intervention
18. Any other condition that the investigator considers would make the participant unsuitable for the clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of OsrHSA on elevating the serum albumin level. | Day 1 to Day 14
  Percentage of participants whose albumin level reaches 35 g/L or above at any time up to 14 days of the study intervention.

SECONDARY OUTCOMES:
To estimate the time to reach 35 g/L or more in serum albumin | Day 1 to Day 14
  Time to reach serum albumin 35 g/L or more by the end of the treatment (EOT)
To estimate the change from baseline in serum albumin | Day 1 to Day 14
  To estimate the change from baseline to the end of treatment (EOT) in serum albumin
To estimate the change from baseline in colloid osmotic pressure | Day 1 to Day 14
  The change from baseline to the end of treatment (EOT) will be measured in Colloid osmotic pressure
To estimate the change from baseline in body weight | Day 1 to Day 14
  The change in body weight will be measured from baseline to the end of treatment (EOT)
To estimate the change from baseline in abdominal circumference, and ascites severity | Day 1 to Day 14
  The change in abdominal circumferences will be measured from baseline to the end of treatment (EOT)
To estimate the change from baseline in ascites severity | Day 1 to Day 14
  The change in ascites severity will be measured from baseline to the end of treatment (EOT)

CONTACTS AND LOCATIONS:
Locations (37):
- China (37):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Youan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Chongqing University Three Gorges Hospital, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Mengchao Hepatobiliary Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Nanfang Hospital, Guangzhou, Guangdong
  - The Third Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Huizhou Central People's Hospital, Huizhou, Guangdong
  - Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Liuzhou Worker's Hospital, Liuchow, Guangxi
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Affiliated Hospital Of Zunyi Medical University, Zunyi, Guizhou
  - The Fourth Affiliated Hospital, Harbin Medical University, Harbin, Heilongjiang
  - Luoyang Central Hospital, Luoyang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Sixth People's Hospital of Zhengzhou, Zhengzhou, Henan
  - Jingzhou Central Hospital, Jingzhou, Hubei
  - TaiHe Hospital, Shiyan, Hubei
  - The Central Hospital of Wuhan, Wuhan, Hubei
  - Wuhan Jinyintan Hospital, Wuhan, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei
  - Yueyang Central Hospital, Yueyang, Hunan
  - The Third People's Hospital of Zhenjiang, Zhenjiang, Jiangsu
  - First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - Yichun People's Hospital, Yichun, Jiangxi
  - Hepatobiliary Hospital Of Jilin, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Sixth People's Hospital of Shenyang, Shenyang, Liaoning
  - The People's Hospital of Qinghai, Xining, Qinghai
  - Shandong Public Health Clinical Center, Jinan, Shandong
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Ruian People's Hospital, Rui’an, Zhejiang
  - The First School of Medicine, School of Information and Engineering, The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No